CLINICAL TRIAL: NCT01458743
Title: A Phase I, Single Center, Open Label, Two Groups Study to Assess the Safety and Pharmacokinetics of Ceftaroline in Healthy Chinese Volunteers Following Single and Multiple Administration of 600 mg Ceftaroline Fosamil as 60-minute Intravenous Infusion Every 12 Hours and as 120-minute Intravenous Infusion Every 8 Hours
Brief Title: Ceftaroline China Pharmacokinetics Study
Acronym: CeftarolineChi
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: D3720C00005
Record Dates: First submitted 2011-09-30; First posted 2011-10-25 (Estimated); Last update posted 2017-09-05 (Actual); Status verified 2017-09

CONDITIONS: Healthy
Keywords: pharmacokinetics
MeSH Terms: interventions — Ceftaroline

ARMS (2):
- Ceftaroline q12h (Experimental): Ceftaroline 600mg q12h
  Interventions: Drug: Ceftaroline
- Ceftaroline q8h (Experimental): ceftaroline 600mg q8h
  Interventions: Drug: Ceftaroline

INTERVENTIONS:
Drug: Ceftaroline — 60-minute single intravenous dose of 600 mg of Ceftaroline on Days 1 and 8; 60-minute intravenous dose of 600 mg of Ceftaroline twice per day on Days 3-7.
  Arms: Ceftaroline q12h
Drug: Ceftaroline — Single intravenous dose on Days 1 and 9. Intravenous three times per day on Days 2-8.
  Arms: Ceftaroline q8h

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics, safety and tolerability of ceftaroline in Chinese healthy subjects following single and multiple intravenous doses.

DETAILED DESCRIPTION:
A Phase I, Single Center and Open Label Study to Assess the Safety and Pharmacokinetics of Ceftaroline in Healthy Chinese Volunteers Following Single and Multiple Administration of 600 mg Ceftaroline Fosamil as 60-minute Intravenous Infusion Every 12 hours and as 120-minute Intravenous Infusion Every 8 hours.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures.
* Are healthy male or female Chinese volunteers aged between 18 and 45 inclusive.
* Have a Body Mass Index (BMI) between (and including) 19 and 24 kg/m2 and weigh at least 50 kg.
* Be willing to communicate with the investigator and comply with all study procedures.

Exclusion Criteria:

* Creatine clearance <80 mL/min as calculated by the Cockcroft Gault equation
* History of any hypersensitivity or allergic reaction to any β-lactam antimicrobial.
* Symptoms of any clinically significant illness within 2 weeks of screening.
* Use of any other investigational compound or participation in another clinical trial within 2 months prior to Visit 2.
* Blood donation with 3 months of screening.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2011-10; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Area under the concentration curve of Ceftaroline over the time (AUC). | Group1: Samples taken on Day 8:Pre-dose, 20 min, 40 min, 55 min, 65 min, 75 min, 1.5 hr, 2 hr, 3 hr ,4 hr, 6hr , 8 hr, 12 hr, 18 hr, 24 hr, 36 hr and 48 hr after the start of infusion of the study drug.
Area under the concentration curve of Ceftaroline over the time (AUC). | Group2: Day3 and Day 5 through 8: pre-dose; Day 4: Pre-dose, 60 min, 90 min, 115 min, 125 min, 2 hr15min, 2.5hr, 3 hr ,4hr, 6hr, 8 hr after the start of infusion of the study drug.
Area under the concentration curve of Ceftaroline over the time (AUC). | Group 2: Day 9: Pre-dose, 60 min, 90 min, 115 min, 125 min, 2 hr15min, 2.5hr, 3 hr ,4 hr, 6hr, 8 hr,12hr,18hr,24hr after the start of infusion of the study drug.
Maximum plasma concentration (Cmax) of Ceftaroline. | Group1: Samples taken on Day 8:Pre-dose, 20 min, 40 min, 55 min, 65 min, 75 min, 1.5 hr, 2 hr, 3 hr ,4 hr, 6hr , 8 hr, 12 hr, 18 hr, 24 hr, 36 hr and 48 hr after the start of infusion of the study drug.
Maximum plasma concentration (Cmax) of Ceftaroline. | Group2:Days 2 through 7: Pre-dose Day 8: Pre-dose, 60 min,90 min,115 min,125 min,2 hr15min,2.5hr,3 hr,4 hr,6hr, 8 hr,12hr,18hr,24hr after the start of infusion of the study drug
Area under the concentration curve of Ceftaroline over the time (AUC) | Group1: Samples taken on Day 1:Pre-dose, 20 min, 40 min, 55 min, 65 min, 75 min, 1.5 hr, 2 hr, 3 hr ,4 hr, 6hr , 8 hr, 12 hr, 18 hr, 24 hr, 36 hr and 48 hr after the start of infusion of the study drug.
Area under the concentration curve of Ceftaroline over the time (AUC) | Group2: Samples taken on Day 1:Pre-dose, 60 min, 90 min, 115 min, 125 min, 2 hr15min, 2.5hr, 3 hr ,4 hr, 6hr , 8 hr, 12 hr, 18 hr, 24 hr after the start of infusion of the study drug.
Maximum plasma concentration (Cmax) of Ceftaroline | Group1: Samples taken on Day 1:Pre-dose, 20 min, 40 min, 55 min, 65 min, 75 min, 1.5 hr, 2 hr, 3 hr ,4 hr, 6hr , 8 hr, 12 hr, 18 hr, 24 hr, 36 hr and 48 hr after the start of infusion of the study drug.
Maximum plasma concentration (Cmax) of Ceftaroline | Group2: Samples taken on Day 1:Pre-dose, 60 min, 90 min, 115 min, 125 min, 2 hr15min, 2.5hr, 3 hr ,4 hr, 6hr , 8 hr, 12 hr, 18 hr, 24 hr after the start of infusion of the study drug.

SECONDARY OUTCOMES:
Area under the concentration curve of Ceftaroline metabolite (Ceftaroline M-1) over the time (AUC). | Group1: Samples taken on Day 1:Pre-dose, 20 min, 40 min, 55 min, 65 min, 75 min, 1.5 hr, 2 hr, 3 hr ,4 hr, 6hr , 8 hr, 12 hr, 18 hr, 24 hr, 36 hr and 48 hr after the start of infusion of the study drug.
Area under the concentration curve of Ceftaroline metabolite (Ceftaroline M-1) over the time (AUC). | Group2: Samples taken on Day 1:Pre-dose, 60 min, 90 min, 115 min, 125 min, 2 hr15min, 2.5hr, 3 hr ,4 hr, 6hr , 8 hr, 12 hr, 18 hr, 24 hr after the start of infusion of the study drug.
Maximum plasma concentration (Cmax) of Ceftaroline metabolite (Ceftaroline M-1) | Group1: Samples taken on Day 1:Pre-dose, 20 min, 40 min, 55 min, 65 min, 75 min, 1.5 hr, 2 hr, 3 hr ,4 hr, 6hr , 8 hr, 12 hr, 18 hr, 24 hr, 36 hr and 48 hr after the start of infusion of the study drug.
Maximum plasma concentration (Cmax) of Ceftaroline metabolite (Ceftaroline M-1) | Group2: Samples taken on Day 1:Pre-dose, 60 min, 90 min, 115 min, 125 min, 2 hr15min, 2.5hr, 3 hr ,4 hr, 6hr , 8 hr, 12 hr, 18 hr, 24 hr after the start of infusion of the study drug.
Area under the concentration curve of Ceftaroline metabolite (Ceftaroline M-1) over the time (AUC). | Group1: Samples taken on Day 8:Pre-dose, 20 min, 40 min, 55 min, 65 min, 75 min, 1.5 hr, 2 hr, 3 hr ,4 hr, 6hr , 8 hr, 12 hr, 18 hr, 24 hr, 36 hr and 48 hr after the start of infusion of the study drug.
Area under the concentration curve of Ceftaroline metabolite (Ceftaroline M-1) over the time (AUC). | Group2:Days 2 through 7:Pre-dose Day8: Pre-dose,60 min,90 min,115 min,125 min, 2 hr 15min,2.5hr,3 hr,4 hr,6hr,8 hr,12hr,18hr,24hr after the start of infusion of the study drug.
Maximum plasma concentration (Cmax) of Ceftaroline metabolite (Ceftaroline M-1) | Group1: Samples taken on Day 8:Pre-dose, 20 min, 40 min, 55 min, 65 min, 75 min, 1.5 hr, 2 hr, 3 hr ,4 hr, 6hr , 8 hr, 12 hr, 18 hr, 24 hr, 36 hr and 48 hr after the start of infusion of the study drug.
Number of patients with adverse events. | From baseline to day 10
Maximum plasma concentration (Cmax) of Ceftaroline metabolite (Ceftaroline M-1) | Group2: Day3 and Day 5 through 8: pre-dose; Day 4: Pre-dose, 60 min, 90 min, 115 min, 125 min, 2 hr 15min, 2.5hr, 3 hr ,4hr, 6hr, 8 hr after the start of infusion of the study drug.
Maximum plasma concentration (Cmax) of Ceftaroline metabolite (Ceftaroline M-1) | Group2: Day 9: Pre-dose, 60 min, 90 min, 115 min, 125 min, 2 hr15min, 2.5hr, 3 hr ,4 hr, 6hr, 8 hr, 12hr, 18hr, 24hr after the start of infusion of the study drug.
Area under the concentration curve of Ceftaroline fosamil over the time (AUC). | Group1: Samples taken on Day 1:Pre-dose, 20 min, 40 min, 55 min, 65 min, 75 min, 1.5 hr, 2 hr, 3 hr ,4 hr, 6hr , 8 hr, 12 hr, 18 hr, 24 hr, 36 hr and 48 hr after the start of infusion of the study drug.
Area under the concentration curve of Ceftaroline fosamil over the time (AUC). | Group2: Samples taken on Day 1:Pre-dose, 60 min, 90 min, 115 min, 125 min, 2 hr15min, 2.5hr, 3 hr ,4 hr, 6hr , 8 hr, 12 hr, 18 hr, 24 hr after the start of infusion of the study drug.
Maximum plasma concentration (Cmax) of Ceftaroline fosamil | Group1: Samples taken on Day 1:Pre-dose, 20 min, 40 min, 55 min, 65 min, 75 min, 1.5 hr, 2 hr, 3 hr ,4 hr, 6hr , 8 hr, 12 hr, 18 hr, 24 hr, 36 hr and 48 hr after the start of infusion of the study drug.
Maximum plasma concentration (Cmax) of Ceftaroline fosamil | Group2: Samples taken on Day 1:Pre-dose, 60 min, 90 min, 115 min, 125 min, 2 hr15min, 2.5hr, 3 hr ,4 hr, 6hr , 8 hr, 12 hr, 18 hr, 24 hr after the start of infusion of the study drug.
Area under the concentration curve of Ceftaroline fosamil over the time (AUC). | Group1: Samples taken on Day 8:Pre-dose, 20 min, 40 min, 55 min, 65 min, 75 min, 1.5 hr, 2 hr, 3 hr ,4 hr, 6hr , 8 hr, 12 hr, 18 hr, 24 hr, 36 hr and 48 hr after the start of infusion of the study drug.
Area under the concentration curve of Ceftaroline fosamil over the time (AUC). | Group2: Day3 and Day 5 through 8: pre-dose; Day 4: Pre-dose, 60 min, 90 min, 115 min, 125 min, 2 hr15min, 2.5hr, 3 hr ,4hr, 6hr, 8 hr after the start of infusion of the study drug.
Area under the concentration curve of Ceftaroline fosamil over the time (AUC). | Group2: Day 9: Pre-dose, 60 min, 90 min, 115 min, 125 min, 2 hr15min, 2.5hr, 3 hr ,4 hr, 6hr, 8 hr,12hr,18hr,24hr after the start of infusion of the study drug.
Maximum plasma concentration (Cmax) of Ceftaroline fosamil | Group1: Samples taken on Day 8:Pre-dose, 20 min, 40 min, 55 min, 65 min, 75 min, 1.5 hr, 2 hr, 3 hr ,4 hr, 6hr , 8 hr, 12 hr, 18 hr, 24 hr, 36 hr and 48 hr after the start of infusion of the study drug.
Maximum plasma concentration (Cmax) of Ceftaroline fosamil | Group2: Day3 and Day 5 through 8: pre-dose; Day 4: Pre-dose, 60 min, 90 min, 115 min, 125 min, 2 hr 15min, 2.5hr, 3 hr ,4hr, 6hr, 8 hr after the start of infusion of the study drug.
Maximum plasma concentration (Cmax) of Ceftaroline fosamil | Group2: Day 9: Pre-dose, 60 min, 90 min, 115 min, 125 min, 2 hr15min, 2.5hr, 3 hr ,4 hr, 6hr, 8 hr,12hr,18hr,24hr after the start of infusion of the study drug.

CONTACTS AND LOCATIONS:
Overall Officials: David Melnick, Study Director — AstraZeneca Pharmaceuticals-US
Locations (1):
- Beijing, China

REFERENCES:
- [Derived] Li J, Das S, Zhou D, Al-Huniti N. Population Pharmacokinetic Modeling and Probability of Target Attainment Analyses in Asian Patients With Community-Acquired Pneumonia Treated With Ceftaroline Fosamil. Clin Pharmacol Drug Dev. 2019 Jul;8(5):682-694. doi: 10.1002/cpdd.673. Epub 2019 May 1. PMID 31044546
- [Derived] Das S, Li J, Iaconis J, Zhou D, Stone GG, Yan JL, Melnick D. Ceftaroline fosamil doses and breakpoints for Staphylococcus aureus in complicated skin and soft tissue infections. J Antimicrob Chemother. 2019 Feb 1;74(2):425-431. doi: 10.1093/jac/dky439. PMID 30380060
- [Derived] Yang L, Sunzel M, Xu P, Edeki T, Wilson D, Li J, Li H. Evaluation of the pharmacokinetics and safety of single and multiple ceftaroline fosamil infusions in healthy Chinese and Western subjects. Int J Clin Pharmacol Ther. 2015 Aug;53(8):681-91. doi: 10.5414/CP202343. PMID 26152131
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=1375&filename=CSR-D3720C00005.pdf
- See also: CSR-D3720C00005.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=1375&filename=CSR-D3720C00005.pdf
- See also: Revised_CSP_1_Redacted_12.03.14 — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1375&filename=D3720C00005_Revised_CSP_1_Redacted_12.03.14.pdf